CLINICAL TRIAL: NCT03055611
Title: A 24-month Prospective, Non-interventional, Multicentre Study to Evaluate the Real-World Usage and Effectiveness of Elocta and Alprolix in Patients With Haemophilia A or B
Brief Title: A Study to Evaluate the Real-world Usage and Effectiveness of Elocta and Alprolix in Patients With Haemophilia A or B
Acronym: PREVENT
Status: Completed | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Other Study IDs: Sobi.HAEM89-002
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Haemophilia A; Haemophilia B
Keywords: Blood Coagulation Disorder; Hematologic Diseases; Coagulation Protein Disorder; Hemorrhagic Disorder; Genetic Diseases, Inborn
MeSH Terms: conditions — Hemophilia A; Hemophilia B; Blood Coagulation Disorders; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn | interventions — factor VIII-Fc fusion protein; factor IX Fc fusion protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Haemophilia A patients: Elocta will be prescribed according to local practice and administered by patients with haemophilia A for prophylactic treatment
  Interventions: Drug: ELOCTA
- Haemophilia B patients: Alprolix will be prescribed according to local practice and administered by patients with haemophilia B for prophylactic treatment
  Interventions: Drug: ALPROLIX

INTERVENTIONS:
Drug: ELOCTA — Extended half-life factor VIII product
  Other Names: Eloctate, efmoroctocog alfa, rFVIIIFc
  Groups: Haemophilia A patients
Drug: ALPROLIX — Extended half-life factor IX product
  Other Names: Eftrenonacog alfa, rFIXFc
  Groups: Haemophilia B patients

SUMMARY:
Elocta (rFVIIIFc) and Alprolix (rFIXFc) are recombinant extended half-life coagulation factor products. The purpose of this non-interventional study is to describe the real-world usage and effectiveness of Elocta and Alprolix in the prophylactic treatment of haemophilia A and B.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of haemophilia A or B and previously treated with factor Product
* Have started prophylactic Elocta/Alprolix treatment prior to enrollment visit, or at enrollment prescribed prophylactic treatment with Elocta or Alprolix regardless of participation in the study
* Signed and dated informed consent provided by the patient, or the patient's legally acceptable representative for patients under the legal age, Before any study-related activities are undertaken. Assent should be obtained from paediatric patients according to local regulations.

Exclusion Criteria:

* Participation in an investigational medicinal product trial, from four weeks prior to first injection with Elocta or Alprolix to enrollment visit.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligible Elocta and Alprolix patients who present for a routine Clinical visit will be asked to participate in the study by the treating physician at participating haemophilia treatment centres in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Annualised bleeding rate (ABR) | 24 months
  Based on bleeding episodes assessed by local practice
Annualised injection frequency | 24 months
  Assessed by prescription
Annualised factor consumption (IU) | 24 months
  Assessed by dispensed factor product

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, MD, Study Director — Swedish Orphan Biovitrum
Locations (22):
- Germany (22):
  - Swedish Orphan Biovitrum Reserach site, Berlin
  - Swedish Orphan Biovitrum Reserach Site, Blaubeuren Abbey
  - Swedish Orphan Biovitrum Research Site, Bonn
  - Swedish Orphan Biovitrum Research Site, Delmenhorst
  - Swedish Orphan Biovitrum Research Site, Duisburg
  - Swedish Orphan Biovitrum Reserach site, Erlangen
  - Swedish Orphan Biovitrum Research Site, Frankfurt
  - Swedish Orphan Biovitrum Reserach site, Frankfurt
  - Swedish Orphan Biovitrum Research Site, Fürth
  - Swedish Orphan Biovitrum Research Site, Hamburg
  - Swedish Orphan Biovitrum Research Site, Hanover
  - Swedish Orphan Biovitrum Reserach site, Hanover
  - Swedish Orphan Biovitrum Reserach site, Heidelberg
  - Swedish Orphan Biovitrum Reserach site, Homburg
  - Swedish Orphan Biovitrum Research Site, Jena
  - Swedish Orphan Biovitrum Reserach Site, Jena
  - Swedish Orphan Biovitrum Reserach site, Leipzig
  - Swedish Orphan Biovitrum Reserach Site, Mörfelden-Walldorf
  - Swedish Orphan Biovitrum Research Site, München
  - Swedish Orphan Biovitrum Reserach site, München
  - Swedish Orphan Biovitrum Reserach site, Münster
  - Swedish Orphan Biovitrum Research Site, Würzburg